CLINICAL TRIAL: NCT02395601
Title: A Phase 1 Study of CPI-1205, a Small Molecule Inhibitor of EZH2, in Patients With B-Cell Lymphomas
Brief Title: A Study Evaluating CPI-1205 in Patients With B-Cell Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Constellation Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1205-01
Record Dates: First submitted 2015-03-10; First posted 2015-03-23 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: B-Cell Lymphoma
Keywords: B-Cell Lymphoma; EZH2 Inhibitor; Phase 1
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — (R)-N-((4-methoxy-6-methyl-2-oxo-1,2-dihydropyridin-3-yl)methyl)-2-methyl-1-(1-(1-(2,2,2-trifluoroethyl)piperidin-4-yl)ethyl)-1H-indole-3-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPI-1205 (Experimental)
  Interventions: Drug: CPI-1205

INTERVENTIONS:
Drug: CPI-1205 — Small molecule inhibitor of the enzyme EZH2

SUMMARY:
First in human, open-label, sequential dose escalation and expansion study of CPI-1205 in patients with progressive B-cell lymphomas. CPI-1205 is a small molecule inhibitor of EZH2.

ELIGIBILITY:
Inclusion Criteria:

Adults (aged ≥ 18 years)

Histologically confirmed diagnosis of a B-cell lymphoma that has progressed in spite of prior treatment, and for which additional effective standard therapy is not available

Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Adequate hematological, renal, hepatic, and coagulation laboratory assessments

Must give written informed consent to participate in this study before the performance of any study-related procedure

Exclusion Criteria:

A primary lymphoma of the central nervous system (CNS) or known lymphomatous involvement of the CNS

Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of CPI-1205, including any unresolved nausea, vomiting, or diarrhea that is CTCAE grade >1

Treatment with proton pump inhibitors, H2 antagonists, or antacids

Achlorhydria, either documented or suspected on the basis of an associated disease (e.g., pernicious anemia, atrophic gastritis, or certain gastric surgical procedures)

Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

* Acute myocardial infarction or angina pectoris ≤ 6 months prior to starting study drug
* New York Heart Association Class III or IV congestive heart failure
* QTcF > 470 msec on the screening ECG

Uncontrolled cardiac arrhythmia (patients with rate-controlled atrial fibrillation are not excluded)

A past medical history of other clinically significant cardiovascular disease (e.g., uncontrolled hypertension, history of labile hypertension or history of poor compliance with an antihypertensive regimen)

Any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study (e.g., clinically significant pulmonary disease, clinically significant neurological disorder, active or uncontrolled infection)

Systemic anti-cancer treatment or radiotherapy less than 2 weeks before the first dose of CPI 1205

Radioimmunotherapy (e.g., 131I-tositumomab, 90Y-ibritumomab tiuxetan) less than 6 weeks before the first dose of CPI-1205

Treatment with an investigational small molecule less than 2 weeks before the first dose of CPI-1205.

Treatment with a therapeutic antibody less than 4 weeks before the first dose of CPI-1205.

Treatment with medications that are strong inhibitors of CYP3A4

Treatment with medications that are inducers of CYP3A4 enzymes

Treatment with medications that are known to carry a risk of Torsades de Pointes

Pregnant or lactating women

Women of child bearing potential and men with reproductive potential, if they are unwilling to use adequate contraception while on study therapy and for 3 months thereafter

Patients unwilling or unable to comply with this study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Dose-limiting toxicities (DLTs) | DLTs asessed during Cycle 1 (first 28 days on study)
  Frequency of dose-limiting toxicities (DLTs) associated with CPI-1205 administration during the first cycle (first 28 days) of treatment

SECONDARY OUTCOMES:
Frequency of adverse events | Assessed from Day 1 of Cycle 1 through 30 days after patient's last dose of study drug
  Safety and tolerability of CPI-1205 as assessed by: frequency of adverse events and serious adverse events; changes in hematology and clinical chemistry values; changes in physical examination, vital signs, electrocardiogram, and ECOG score
Pharmacokinetic parameters of CPI-1205: AUC(0-t), AUC(0-inf), AUCtau,ss, Tmax, Cmax, Ctrough, T1/2, Vd/F, CL/F | Assessed during cycle 1 (first 28 days on study); and on cycle 2, day 1
Pharmacodynamic effects of CPI-1205 in lymphoma tissue: changes in levels of the trimethylated form of lysine residue 27 on histone 3; changes in the expression of genes whose transcription may be altered by EZH2 inhibition | Assessed during cycle 1 (first 28 days on study)
Pharmacodynamic effects of CPI-1205 in bone marrow and in skin: changes in global levels of the trimethylated form of lysine residue 27 on histone 3 (H3K27me3) | Assessed during cycle 1 (first 28 days on study)
Disease response assessment will be performed using the 2014 Lugano Response Criteria for Hodgkin and Non-Hodgkin Lymphoma | After every 2 cycles of treatment for the first 6 cycles, and after every 4 cycles thereafter

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Horizon Oncology Center, Lafayette, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - John Theurer Cancer Center, Hackensack, New Jersey
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee